CLINICAL TRIAL: NCT02483429
Title: Acute Video-oculography for Vertigo in Emergency Rooms for Rapid Triage (AVERT)
Acronym: AVERT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); GN Otometrics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00044228; 1U01DC013778-01A1 (NIH)
Record Dates: First submitted 2015-03-03; First posted 2015-06-29 (Estimated); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Vertigo; Dizziness
Keywords: Vertigo; Dizziness; Unsteadiness; Stroke; Vestibular neuritis; Benign paroxysmal positional vertigo; Vestibulo-ocular reflex; Video-oculography; Emergency department
MeSH Terms: conditions — Vertigo; Dizziness; Stroke; Vestibular Neuronitis; Benign Paroxysmal Positional Vertigo; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- VRT Care (Experimental): Patients randomized to VRT (VOG-guided Rapid Triage) care will have an algorithm-determined patient-specific diagnosis and treatment pathway in the emergency department. Participants will complete a 1-week in-person follow-up and a 1-month and 6-month phone follow-up.
  Interventions: Device: VRT Care
- Standard of Care (SOC) (No Intervention): Patients randomized to Standard of Care will undergo usual emergency department care without revealing results of VOG testing. Participants will complete a 1-week in-person follow-up and a 1-month and 6-month phone follow-up.

INTERVENTIONS:
Device: VRT Care — The VOG report includes direct device output (physiologic traces, quantitative measures) plus most likely diagnosis, category, and clinical trial care pathway (peripheral, equivocal, central) instructions. The VOG report becomes part of the patient's emergency department clinical record.
  Other Names: GN Otometrics (Instrumentation & Control Systems, Inc)
  Arms: VRT Care

SUMMARY:
AVERT is a randomized controlled trial comparing video-oculography (VOG)-guided care to standard care to assess accuracy of diagnoses and initial management decisions for emergency department (ED) patients with a chief symptom of vertigo or dizziness suspected to be of vestibular cause. The trial will test the hypothesis that VOG-guided rapid triage (VRT) will accurately, safely, and efficiently differentiate peripheral from central vestibular disorders in ED patients presenting acute vertigo or dizziness, and that doing so has the potential to improve post-treatment clinical outcomes for these patients.

DETAILED DESCRIPTION:
AVERT is a multicenter phase 2 clinical trial comparing a novel diagnostic strategy (VRT) to standard ED diagnostic care at three performance sites. The Specific Aims are to assess diagnostic accuracy, diagnostic workup costs, and estimate the short-term impact of correct diagnosis in anticipation of a larger, definitive phase 3 trial. Adult ED patients with a chief symptom of vertigo, dizziness, or unsteadiness, new or clearly worse in the previous 30 days, will undergo on-site vestibular function tests by trained research personnel using a portable, quantitative VOG recording device. Research personnel will also record a focused symptom history and bedside hearing tests. Eligible patients with at least one pathologic vestibular eye movement finding or pathologic ataxia will be randomized to VRT or standard ED care. Patients eligible for pre-randomization testing but excluded from randomization will be slated for the Observational Arm of the study and will undergo limited 1-month and 6-month phone follow-up. The VRT arm relies on an automated algorithm to interpret VOG results, thereby determining a patient-specific clinical care pathway. For safety, all VRT-arm study participants will undergo stroke protocol MRI before release. All randomized participants will undergo confirmatory testing at one week, including vestibular specialist exam and 1.5 or 3-Tesla research MRI combining stroke and internal auditory canal protocols. All randomized participants will also undergo 1-month and 6-month phone follow-up and medical record review to confirm diagnoses. Clinical findings, ED diagnoses, diagnostic resource utilization, treatments applied, and clinical events during follow-up will be recorded. A multidisciplinary, masked expert panel will adjudicate final diagnoses.

ELIGIBILITY:
Inclusion criteria:

Adult (18 years and older) ED patients with all of the following (all determined pre-randomization):

* VESTIBULAR SYMPTOMS: presenting symptom of "vertigo" OR "dizziness" OR "unsteadiness" (as defined by consensus expert definitions in the International Classification of Vestibular Disorders).
* RELEVANT EXAM SIGNS*: pathologic nystagmus (spontaneous, gaze-evoked, or positional) by bedside VOG testing OR pathologic ataxia (gait, trunk, stance, limbs) by bedside ataxia examination.
* RECENT ONSET: symptoms AND signs* appear to be new or markedly worse in the past month. (*Exam signs are required for randomization, but not for the observational arm)

Exclusion Criteria

1. Excluded from Pre-Randomization Screening

   * Level 1 trauma or critical illness
   * Altered mental status (e.g., delirium, dementia) that would preclude active study participation (this includes patients with abnormal mental state due to alcohol intoxication or illicit substance, which are known, easily-recognized causes of dizziness or vertigo presentations to the ED)
   * Non-English speaking (enrollment of non-English speakers is not feasible given the logistics of identifying a translator and the need for rapid recruitment and randomization in the AVERT study; furthermore, the terms vertigo, dizziness, and unsteadiness may have different meanings in other languages)
   * Known pregnancy (all women of childbearing age who are enrolled will undergo a urine or serum beta human chorionic gonadotropin [hCG] pregnancy test prior to MRI to confirm no pregnancy, per local institutional guidelines)
   * Unable or unsafe to participate in screening, including VOG tests (as deemed by specific pre-enrollment risk assessment questions or ED provider and/or Study Coordinator judgment) including, but not limited to:

     * visual impairment sufficient to prevent visual fixation during the VOG testing
     * clinically-perceived risk to patient of participating in study (ED provider or staff concerns)
     * clinically-perceived risk to research staff (e.g., violence, blood/body fluid/respiratory precautions)
     * unstable cardiac status (given a single reported case of bradycardia with impulse testing)
     * acute cranio-cervical trauma or other condition (e.g., rheumatoid arthritis) that might lead to instability of the cervical spine that would be a contraindication to neck rotation during VOG testing
   * Obvious general medical cause (as judged by treating ED provider) including, but not limited to, acute myocardial infarction, pulmonary embolus, pneumonia, urinary tract infection, drug intoxication, etc.
2. Excluded from Randomization (Eligible for Observational Arm Follow-up)

   * Patient previously randomized in the AVERT Trial (previously screened but not randomized are eligible)
   * Unable to participate fully with study follow-up (particularly MRI) including, but not limited to:

     * unable to return for follow-up testing within 30 days
     * unable to undergo MRI because of contraindications (e.g., pacemaker, metallic foreign body, pregnancy) or other reasons (severe claustrophobia, too large or too heavy for MRI scanner)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Newman-Toker, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - University of Illinois, Peoria, Illinois
  - Johns Hopkins Hospital - Bayview, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mt. Sinai Medical Center, New York, New York

REFERENCES:
- [Derived] Edlow JA, Carpenter C, Akhter M, Khoujah D, Marcolini E, Meurer WJ, Morrill D, Naples JG, Ohle R, Omron R, Sharif S, Siket M, Upadhye S, E Silva LOJ, Sundberg E, Tartt K, Vanni S, Newman-Toker DE, Bellolio F. Guidelines for reasonable and appropriate care in the emergency department 3 (GRACE-3): Acute dizziness and vertigo in the emergency department. Acad Emerg Med. 2023 May;30(5):442-486. doi: 10.1111/acem.14728. PMID 37166022
- [Derived] Kotwal S, Fanai M, Fu W, Wang Z, Bery AK, Omron R, Tevzadze N, Gold D, Garibaldi BT, Wright SM, Newman-Toker DE. Real-world virtual patient simulation to improve diagnostic performance through deliberate practice: a prospective quasi-experimental study. Diagnosis (Berl). 2021 Mar 8;8(4):489-496. doi: 10.1515/dx-2020-0127. Print 2021 Nov 25. PMID 33675203
- See also: Brain Injury OutcomeS (BIOS) website — http://braininjuryoutcomes.com

RESULTS

PARTICIPANT FLOW:
Groups:
- VRT Care: Patients randomized to video-oculography (VOG)-guided rapid triage (VRT) care will have an algorithm-determined patient-specific diagnosis and treatment pathway in the emergency department (ED). Participants will complete a 1-week in-person follow-up and a 1-month and 6-month phone follow-up.
  VRT Care: The VOG report includes direct device output (physiologic traces, quantitative measures) plus most likely diagnosis, category, and clinical trial care pathway (peripheral, equivocal, central) instructions. The VOG report becomes part of the patient's emergency department clinical record.
Period: Overall Study
Arm/Group | VRT Care | Standard of Care (SOC)
Started | 65 | 65
Completed | 57 | 56
Not Completed | 8 | 9
Not completed — Incomplete 1-week follow-up (excluded from primary analysis) | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRT Care | Standard of Care (SOC) | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (15.8) | 60.1 (14.3) | 59.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 29 | 33 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 60 | 63 | 123
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 10 | 19
  White | 48 | 52 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 65 | 130

OUTCOME MEASURES:

1. Primary Outcome: VRT vs. ED SOC Six-Category Diagnosis Accuracy (Primary Analysis-eligible Participants, Two-arm Comparison)
Description: Total diagnosis accuracy VRT vs. ED SOC using 30-day adjudicated final diagnoses categorized in one of six diagnosis categories (3 peripheral, 1 central, 1 medical/other, 1 non-diagnosis). VRT diagnoses were based on automated interpretation of ED index VOG tests in the context of structured medical history information and examination findings from the ED index visit (clinically supervised for safety), while ED SOC diagnoses were based on all clinical information from the ED index visit, including neuroimaging and consultations. Final diagnoses were based on ED index visit, 1-week, and 30-day follow-up clinical assessments. The population was limited to those with complete 1-week follow-up testing including in-person vestibular specialist exam, repeat VOG assessment, and MRI with diffusion-weighted images for ischemic stroke detection.
Time Frame: 30-day follow-up time point
Population: Randomized participants (n=130) who had complete 1-week follow-up testing (n=113) that included, at a minimum, in-person vestibular specialist exam, repeat VOG assessment, and MRI with diffusion-weighted images for ischemic stroke detection.
Measure: Count of Participants; unit: Participants
Groups:
- VOG-guided Rapid Triage (VRT) Care: Participants in both trial arms underwent video-oculography (VOG) testing to analyze their eye movements and were then randomized either to have VOG results algorithmically analyzed in real time and incorporated into their emergency department (ED) care process or for the VOG results not to be analyzed until a later date (i.e., during the trial's delayed diagnosis adjudication procedures). Participants completed a 1-week in-person follow-up, a 1-month phone follow-up, and a 1-month medical record review. Those completing the required 1-week follow-up testing (in-person vestibular specialist examination, repeat VOG testing, and follow-up MRI for ischemic stroke detection) were eligible for the primary analysis of the main trial outcomes as prespecified in the AVERT protocol at the trial's outset.
  VRT Care: Participants randomized to VRT (VOG-guided Rapid Triage) care received an automated algorithm-determined, patient-specific diagnosis and treatment pathway in the ED based on VOG testing. Automated algorithm outputs were reviewed for safety by an on-call trial physician before being incorporated into the patient's ED care process. The VOG report included direct device output (physiologic traces, quantitative measures) plus an algorithmically generated most likely diagnosis, diagnosis category (peripheral, equivocal, central), and diagnosis-specific clinical trial care pathway instructions. The VOG report was incorporated into the patient's ED care and clinical record.
- Standard of Care (SOC) Care: Participants in both trial arms underwent video-oculography (VOG) testing to analyze their eye movements and were then randomized either to have VOG results algorithmically analyzed in real time and incorporated into their emergency department (ED) care process or for the VOG results not to be analyzed until a later date (i.e., during the trial's delayed diagnosis adjudication procedures). Participants completed a 1-week in-person follow-up, a 1-month phone follow-up, and a 1-month medical record review. Those completing the required 1-week follow-up testing (in-person vestibular specialist examination, repeat VOG testing, and follow-up MRI for ischemic stroke detection) were eligible for the primary analysis of the main trial outcomes as prespecified in the AVERT protocol at the trial's outset.
  SOC Care: Participants randomized to SOC (Standard of Care) care received usual ED care without VOG test results or interpretations being revealed to the ED care team. ED SOC diagnoses were based on all clinical information from the ED index visit, including neuroimaging and consultations.
Arm/Group | VOG-guided Rapid Triage (VRT) Care | Standard of Care (SOC) Care
Number analyzed (Participants) | 57 | 56
Participants
  Participants with a correct ED index visit diagnosis | 24 | 18
  Participants with an incorrect ED index visit diagnosis | 33 | 38

2. Primary Outcome: VRT vs. ED SOC Total Diagnostic Utilization Costs at the ED Index Visit (Primary Analysis-eligible Participants, Two-arm Comparison)
Description: Total US dollar costs VRT vs. ED SOC for diagnostic tests and consultations obtained during the ED index visit and associated hospital admission (for those admitted at the index visit). For the VRT arm, this does not include costs of safety MRIs required by the institutional review board (IRB)-approved protocol or any tests ordered "off protocol" by ED physicians (i.e., it represents VRT-recommended utilization-based costs); however, it does include tests, consultations, or admissions ordered "on protocol" by consultants or ED physicians in the VRT "equivocal" diagnosis pathway. For the SOC arm, this includes all utilization-related costs from the ED index visit (tests, consultations, or admissions). Total costs are calculated by multiplying fixed cost estimates (2025 national average Medicare reimbursement in US dollars) by utilization rates for each ED index visit service tracked.
Time Frame: 30-day follow-up time point
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: US dollars
Arm/Group | VOG-guided Rapid Triage (VRT) Care | Standard of Care (SOC) Care
Number analyzed (Participants) | 57 | 56
US dollars | 3007.1 [2367.9 to 3646.3] | 3599.0 [2986.1 to 4211.8]

3. Primary Outcome: Participants With Short-Term Prespecified Medical Event(s) of Interest (PMEIs) After a Correct vs. Incorrect Diagnosis (Primary Analysis-eligible Participants, One-arm Comparison [SOC Arm Only])
Description: PMEIs included ED revisits, falls, vascular events, and test or treatment complications. PMEIs occurring between the ED index visit disposition and 1-week follow-up visit (after which the two arms joined the same diagnostic pathway) were considered. Events diagnosed at ED index visit were not counted. Events newly diagnosed at 1-week follow-up or in the interval prior to 1-week follow-up were counted, regardless of relatedness to ED index dizziness symptoms, with the exception of test or treatment complications, which were required to be related directly or indirectly to the dizziness symptoms. To avoid "double counting" misdiagnoses as follow-on PMEIs pursuant to an initial misdiagnosis, 1-week stroke diagnoses not rendered at the ED index visit were not counted unless neurologic or vestibular symptoms/signs worsened after the ED index visit. Six-category accuracy was used to determine "correct" vs. "incorrect" index ED SOC diagnoses relative to 30-day adjudicated final diagnoses.
Time Frame: 1-week follow-up time point
Population: Randomized participants in the SOC Care trial arm (n=65) who had complete 1-week follow-up testing (n=56) that included, at a minimum, in-person vestibular specialist exam, repeat VOG assessment, and MRI with diffusion-weighted images for ischemic stroke detection.
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care (SOC) Care Trial Arm Participants With a Correct ED SOC Diagnosis: SOC Care: Participants randomized to SOC (Standard of Care) care received usual ED care without VOG test results or interpretations being revealed to the ED care team. ED SOC diagnoses were based on all clinical information from the ED index visit, including neuroimaging and consultations.
  Correctness of ED SOC index visit diagnosis: Participants with ED SOC index visit diagnoses matching the six-category, 30-day adjudicated final diagnosis were considered "correct."
- Standard of Care (SOC) Care Trial Arm Participants With an Incorrect ED SOC Diagnosis: SOC Care: Participants randomized to SOC (Standard of Care) care received usual ED care without VOG test results or interpretations being revealed to the ED care team. ED SOC diagnoses were based on all clinical information from the ED index visit, including neuroimaging and consultations.
  Correctness of ED SOC index visit diagnosis: Participants with ED SOC index visit diagnoses NOT matching the six-category, 30-day adjudicated final diagnosis were considered "incorrect."
Arm/Group | Standard of Care (SOC) Care Trial Arm Participants With a Correct ED SOC Diagnosis | Standard of Care (SOC) Care Trial Arm Participants With an Incorrect ED SOC Diagnosis
Number analyzed (Participants) | 18 | 38
Participants
  Participants with zero PMEIs | 17 | 35
  Participants with one or more PMEIs | 1 | 3

4. Secondary Outcome: Expert VOG vs. ED SOC Six-Category Diagnosis Accuracy (Participants With a Known Final Diagnosis, One-arm Comparison [SOC Arm Only])
Description: Total diagnosis accuracy Expert VOG vs. ED SOC using 30-day adjudicated final diagnoses categorized in one of six diagnosis categories (3 peripheral, 1 central, 1 medical/other, 1 non-diagnosis). Expert VOG diagnoses were based on masked interpretation of ED index VOG tests in the context of basic demographic and medical history information from the ED index visit, while ED SOC diagnoses were based on all clinical information from the ED index visit, including neuroimaging and consultations. Final diagnoses were based on ED index visit, 1-week, and 30-day follow-up clinical assessments. The SOC arm population was limited to those with known final diagnoses to avoid counting as "incorrect" cases with unknown final diagnoses after 30-day follow-up. This within-subject comparison reflects current potential accuracy of expert VOG-based tele-diagnosis and the targeted maximum diagnostic accuracy (i.e., expert level performance) for future automated algorithms, relative to current care.
Time Frame: 30-day follow-up time point
Population: Randomized participants in the SOC Care trial arm (n=65) who had a known final diagnosis (n=51).
Measure: Count of Participants; unit: Participants
Groups:
- Expert VOG Diagnosis Within SOC Care Trial Arm: SOC Care: Participants randomized to SOC (Standard of Care) care received usual ED care without VOG test results or interpretations being revealed to the ED care team.
  Expert VOG Diagnosis: Expert VOG diagnoses were based on masked interpretation of ED index visit VOG tests accompanied by basic demographic and medical history information, as would be available in a routine tele-consultation. This assessment was performed by vestibular specialists as a component of the diagnosis adjudication process and was masked to all other clinical data including ED index visit neuroimaging, consultation, and final ED index disposition as well as all follow-up data occurring after the ED index visit.
- ED SOC Diagnosis Within SOC Care Trial Arm: SOC Care: Participants randomized to SOC (Standard of Care) care received usual ED care without VOG test results or interpretations being revealed to the ED care team.
  ED SOC Diagnoses: ED SOC diagnoses were based on all clinical information from the ED index visit, including any neuroimaging or consultations ordered clinically during the ED index visit. These diagnoses were the final clinical diagnoses rendered in the ED.
Arm/Group | Expert VOG Diagnosis Within SOC Care Trial Arm | ED SOC Diagnosis Within SOC Care Trial Arm
Number analyzed (Participants) | 51 | 51
Participants
  Participants with a correct ED index visit diagnosis | 29 | 13
  Participants with an incorrect ED index visit diagnosis | 22 | 38

5. Secondary Outcome: VRT vs. ED SOC Stroke-No Stroke Diagnosis Accuracy (Primary Analysis-eligible Participants, Two-arm Comparison)
Description: Total diagnosis accuracy VRT vs. ED SOC using 30-day adjudicated final diagnoses categorized as stroke (any cerebrovascular event) versus no stroke (including peripheral vestibular, medical, psychiatric, or other central neurologic causes such as multiple sclerosis, traumatic brain injury, epilepsy, or anticonvulsant toxicity). "Index VRT Diagnosis" and "ED SOC Diagnosis" were compared to the "Adjudicated Final Diagnosis" based on ED index visit and 30-day follow-up clinical assessments.
Time Frame: 30-day follow-up time point
Population: Randomized participants (n=130) who had complete 1-week follow-up testing (n=113) that included, at a minimum, in-person vestibular specialist exam, repeat VOG assessment, and MRI with diffusion-weighted images for ischemic stroke detection. Participants were also required to have a known final stroke diagnosis (n=100).
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care (SOC) Care: Participants in both trial arms underwent video-oculography (VOG) testing to analyze their eye movements and were then randomized either to have VOG results algorithmically analyzed in real time and incorporated into their emergency department (ED) care process or for the VOG results not to be analyzed until a later date (i.e., during the trial's delayed diagnosis adjudication procedures). Participants completed a 1-week in-person follow-up, a 1-month phone follow-up, and a 1-month medical record review. Those completing the required 1-week follow-up testing (in-person vestibular specialist examination, repeat VOG testing, and follow-up MRI for ischemic stroke detection) were eligible for the primary analysis of the main trial outcomes as prespecified in the AVERT protocol at the trial's outset.
  SOC Care: Participants randomized to SOC (Standard of Care) care received usual ED care without VOG test results or interpretations being revealed to the ED care team.
Arm/Group | VOG-guided Rapid Triage (VRT) Care | Standard of Care (SOC) Care
Number analyzed (Participants) | 54 | 46
Participants
  Strokes: Participants with a correct ED index visit diagnosis: number analyzed (Participants) | 8 | 6
  Strokes: Participants with a correct ED index visit diagnosis | 5 | 4
  Strokes: Participants with an incorrect ED index visit diagnosis: number analyzed (Participants) | 8 | 6
  Strokes: Participants with an incorrect ED index visit diagnosis | 3 | 2
  Non-strokes: Participants with a correct ED index visit diagnosis: number analyzed (Participants) | 46 | 40
  Non-strokes: Participants with a correct ED index visit diagnosis | 35 | 39
  Non-strokes: Participants with an incorrect ED index visit diagnosis: number analyzed (Participants) | 46 | 40
  Non-strokes: Participants with an incorrect ED index visit diagnosis | 11 | 1

ADVERSE EVENTS:
Time Frame: Up to 30 days follow-up
Description: Events were assessed systematically during the ED index visit, 1-week follow-up visit, and 1-month follow-up call, and via medical record review. Events associated with VOG testing, as well as any reported test-related adverse events, were systematically tracked throughout the trial.
Arm/Group | VRT Care | Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 47/65 | 53/65
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VRT Care (N=65) | Standard of Care (SOC) (N=65)
Transient increased dizziness, nausea, or vomiting during or immediately after VOG testing (Injury, poisoning and procedural complications) | 40 | 37
Persistent increase in dizziness, nausea, vomiting, or gait unsteadiness after VOG testing (Injury, poisoning and procedural complications) | 7 | 11
Transient fatigue or malaise during or immediately after VOG testing (Injury, poisoning and procedural complications) | 8 | 13
Transient neck discomfort during or immediately after VOG testing (Injury, poisoning and procedural complications) | 7 | 11
Transient discomfort where the goggles sit or mild headache during or immediately after VOG testing (Injury, poisoning and procedural complications) | 20 | 17
Mild skin irritation (including eyelid) from sticky eyepatch or goggles foam insert for VOG testing (Injury, poisoning and procedural complications) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Informed Consent Form: Protocol with sample consent form (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT02483429/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT02483429/SAP_002.pdf
  • Informed Consent Form: Johns Hopkins site informed consent form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT02483429/ICF_003.pdf